CLINICAL TRIAL: NCT01767376
Title: Immunogenicity, Safety and Reactogenicity Study of GSK Biologicals' Meningococcal Conjugate Vaccine (GSK134612) When Co-administered With Boostrix® in Healthy Adolescents and Young Adults Between 11 and 25 Years of Age
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Meningococcal Conjugate Vaccine (GSK134612) When Co-administered With Boostrix® in Subjects Between 11 and 25 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 116705; 2012-002737-11 (EudraCT Number)
Record Dates: First submitted 2012-12-21; First posted 2013-01-14 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Infections, Meningococcal
Keywords: Young adults; Adolescents; Reactogenicity; Diphtheria; pertussis; Immunogenicity; Tetanus; Meningococcal vaccines; Safety; Neisseria meningitidis; Healthy
MeSH Terms: conditions — Meningococcal Infections; Diphtheria; Whooping Cough; Tetanus | interventions — tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine; Boostrix

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Nimenrix+ Boostrix Group (Experimental): Healthy male or female subjects, between and including 11 and 25 years of age, who received one dose of Nimenrix vaccine co-administered with one dose of Boostrix vaccine, at Month 0, administered by intramuscular injection into the deltoid muscle.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Boostrix®
- Nimenrix Group (Experimental): Healthy male or female subjects, between and including 11 and 25 years of age, who received one dose of Nimenrix vaccine at Month 0 and one dose of Boostrix vaccine at Month 1. Both vaccines were administered by intramuscular injection into the deltoid muscle.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Boostrix®
- Boostrix Group (Experimental): Healthy male or female subjects, between and including 11 and 25 years of age, who received one dose of Boostrix vaccine at Month 0 and one dose of Nimenrix vaccine at Month 1. Both vaccines were administered by intramuscular injection into the deltoid muscle.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Boostrix®

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One dose administered intramuscularly (IM) in the deltoid muscle of the arm.
  Other Names: MenACWY-TT; Nimenrix
Biological: Boostrix® — One dose administered intramuscularly (IM) in the deltoid of the right arm (in Co-ad Group) and left arm (in TdapACWY and ACWYTdap Groups).
  Other Names: Tdap

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety and reactogenicity of the meningococcal conjugate vaccine (MenACWY-TT) co-administered with Boostrix® versus each of the two vaccines given separately in healthy adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects and subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 11 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/from the parent(s)/LAR(s) of the subject.
* Written informed assent obtained from the subjects when applicable according to local regulations.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy or ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥ 10 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose of vaccine and ending 30 days after the last dose of vaccine, with the exception of licensed inactivated influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination with a meningococcal vaccine.
* History of meningococcal disease.
* Vaccination with a DTP-containing vaccine within the previous five years.
* History of serious allergic reaction following any other DTP-containing vaccine or any component of the study vaccines.
* History of encephalopathy within seven days following administration of a previous dose of pertussis vaccine that is not attributable to another identifiable cause.
* Temperature of ≥ 40.5°C (105°F) within 48 hours of receipt of a previous dose of DTP vaccine, not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of receipt of a previous dose of DTP vaccine.
* Seizures with or without fever within three days of a previous dose of DTP vaccine.
* Severe Arthus-type hypersensitivity reactions following a prior dose of tetanus toxoid (TT) within the previous ten years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination during the study period.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Progressive neurologic disorder, uncontrolled epilepsy or progressive encephalopathy.
* History of any neurologic disorders or seizures, including Guillain-Barré syndrome (GBS). History of a simple, single febrile seizure is permitted.
* Bleeding disorders, such as haemophilia or thrombocytopenia, or subjects on anticoagulant therapy.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine, or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 692 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2014-01-16 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- GSK Investigational Site, Santo Domingo, Distrito Nacional, Dominican Republic
- Germany (7):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
- South Korea (4):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Seoul

REFERENCES:
- [Derived] Rivera L, Schwarz TF, Kim KH, Kim YK, Behre U, Cha SH, Jo DS, Lee J, Lee JS, Cheuvart B, Jastorff A, Van der Wielen M. Immunogenicity and safety of the quadrivalent meningococcal vaccine MenACWY-TT co-administered with a combined diphtheria-tetanus-acellular pertussis vaccine versus their separate administration in adolescents and young adults: A phase III, randomized study. Vaccine. 2018 Jul 25;36(31):4750-4758. doi: 10.1016/j.vaccine.2018.04.034. Epub 2018 Jun 28. PMID 29960800

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms. Out of the 692 subjects enrolled in this study, one subject was eliminated due to not receiving vaccination, hence only 691 subject started the study.
Period: Overall Study
Arm/Group | Nimenrix+ Boostrix Group | Nimenrix Group | Boostrix Group
Started | 231 | 228 | 232
Completed | 227 | 225 | 232
Not Completed | 4 | 3 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix+ Boostrix Group | Nimenrix Group | Boostrix Group | Total
Number analyzed (Participants) | 231 | 228 | 232 | 691
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.1 (4.2) | 18.2 (4.5) | 18.3 (4.4) | 18.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 126 | 146 | 400
  Male | 103 | 102 | 86 | 291
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian - East Asian Heritage | 111 | 109 | 111 | 331
  Ethnicity: Asian - South East Asian Heritage | 0 | 0 | 1 | 1
  Ethnicity: White - Caucasian / European Heritage | 60 | 60 | 61 | 181
  Ethnicity: Other | 60 | 59 | 59 | 178

OUTCOME MEASURES:

1. Primary Outcome: Anti-Meningitis Antibody Titers by Serum Bactericidal Assay Using Rabbit Complement (rSBA)
Description: The analysis was performed for the serogroups -MenA, -MenC -MenW-135 and -MenY. Antibody titers tabulated as geometric mean titers (GMTs), were obtained by serum bactericidal assay using rabbit complement and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL). The primary outcome results only refer to Nimenrix+Boostrix Group and Nimenrix Group.
Time Frame: One month after Nimenrix vaccination (i.e. Month 1 for Nimenrix+Boostrix and Nimenrix Groups and Month 2 for Boostrix Group)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity will included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component after at least one vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Nimenrix + Boostrix Group: Healthy male or female subjects, between and including 11 and 25 years of age, who received one dose of Nimenrix vaccine co-administered with one dose of Boostrix vaccine, at Month 0, administered by intramuscular injection into the deltoid muscle.
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 226 | 222 | 223
EL.U/mL
  rSBA-MenA: number analyzed (Participants) | 225 | 222 | 223
  rSBA-MenA | 3415.3 [2917.8 to 3997.6] | 2860.4 [2478.6 to 3300.9] | 1577.4 [1354.4 to 1837.1]
  rSBA-MenC | 5092.5 [4268.7 to 6075.3] | 4597.6 [3703.1 to 5708.2] | 1912.6 [1593.9 to 2295.1]
  rSBA-MenW-135 | 9608.5 [8522.5 to 10832.8] | 9052.8 [7510.3 to 10912.0] | 3164.6 [2534.0 to 3952.1]
  rSBA-MenY | 7775.8 [6862.3 to 8811.0] | 6032.6 [5025.7 to 7241.2] | 4134.4 [3582.3 to 4771.5]
Statistical Analysis 1: Comparison: Nimenrix + Boostrix Group vs Nimenrix Group; To demonstrate the non-inferiority of Nimenrix co-administered with Boostrix (Nimenrix+Boostrix Group) compared to Nimenrix administered alone (Nimenrix Group) with respect to serum bactericidal assay using rabbit complement (rSBA) geometric mean titers (GMTs) for serogroup A, one month after Nimenrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardised asymptotic 95% confidence interval (CI) for rSBA GMT ratios for serogroup A between the two groups (Nimenrix+Boostrix Group minus Nimenrix Group) being greater than or equal to (≥) the pre-defined limit of 0.5; ANCOVA; Adjusted GMT ratio = 1.19, 95% CI 2-sided [0.97 to 1.48]
Statistical Analysis 2: Comparison: Nimenrix + Boostrix Group vs Nimenrix Group; To demonstrate the non-inferiority of Nimenrix co-administered with Boostrix (Nimenrix+Boostrix Group) compared to Nimenrix administered alone (Nimenrix Group) with respect to serum bactericidal assay using rabbit complement (rSBA) geometric mean titers (GMTs) for serogroup C, one month after Nimenrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardised asymptotic 95% confidence interval (CI) for rSBA GMT ratios for serogroup C between the two groups (Nimenrix+Boostrix Group minus Nimenrix Group) being greater than or equal to (≥) the pre-defined limit of 0.5; ANCOVA; Adjusted GMT ratio = 1.12, 95% CI 2-sided [0.85 to 1.47]
Statistical Analysis 3: Comparison: Nimenrix + Boostrix Group vs Nimenrix Group; To demonstrate the non-inferiority of Nimenrix co-administered with Boostrix (Nimenrix+Boostrix Group) compared to Nimenrix administered alone (Nimenrix Group) with respect to serum bactericidal assay using rabbit complement (rSBA) geometric mean titers (GMTs) for serogroup W-135, one month after Nimenrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardised asymptotic 95% confidence interval (CI) for rSBA GMT ratios for serogroup W-135 between the two groups (Nimenrix+Boostrix Group minus Nimenrix Group) being greater than or equal to (≥) the pre-defined limit of 0.5; ANCOVA; Adjusted GMT ratio = 1.06, 95% CI 2-sided [0.86 to 1.32]
Statistical Analysis 4: Comparison: Nimenrix + Boostrix Group vs Nimenrix Group; To demonstrate the non-inferiority of Nimenrix co-administered with Boostrix (Nimenrix+Boostrix Group) compared to Nimenrix administered alone (Nimenrix Group) with respect to serum bactericidal assay using rabbit complement (rSBA) geometric mean titers (GMTs) for serogroup Y, one month after Nimenrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardised asymptotic 95% confidence interval (CI) for rSBA GMT ratios for serogroup Y between the two groups (Nimenrix+Boostrix Group minus Nimenrix Group) being greater than or equal to (≥) the pre-defined limit of 0.5; ANCOVA; Adjusted GMT ratio = 1.27, 95% CI 2-sided [1.02 to 1.59]

2. Primary Outcome: Number of Subjects With Anti-D and Anti-T Concentrations Above the Cut-off Value
Description: The antibody concentrations were calculated as geometric mean concentrations (GMCs) and expressed as international units per milliliter (IU/mL). The reference cut-off value was an antibody concentration ≥ 1 IU/mL. The primary outcome results only refer to Nimenrix+Boostrix Group and Boostrix Group.
Time Frame: One month after Boostrix vaccination (i.e. Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity will included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component after at least one vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Boostrix Group
Number analyzed (Participants) | 225 | 223
Participants
  Anti-D | 200 | 203
  Anti-T | 224 | 223
Statistical Analysis 1: Comparison: Nimenrix + Boostrix Group vs Boostrix Group; To demonstrate the non-inferiority of Boostrix co-administered with Nimenrix (Nimenrix+Boostrix Group) compared to Boostrix administered alone (Boostrix Group) in terms of anti-diphtheria toxoid (anti-D) antibody concentrations one month after Boostrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) between the two groups (Nimenrix+Boostrix Group minus Boostrix Group), in terms of percentage of subjects with anti-D concentrations ≥ 1.0 IU/mL, being greater than or equal to (≥) the pre-defined limit of -10%; Difference in percentage = -2.14, 95% CI 2-sided [-7.88 to 3.53]
Statistical Analysis 2: Comparison: Nimenrix + Boostrix Group vs Boostrix Group; To demonstrate the non-inferiority of Boostrix co-administered with Nimenrix (Nimenrix+Boostrix Group) compared to Boostrix administered alone (Boostrix Group) in terms of anti-tetanus toxoid (anti-T) antibody concentrations one month after Boostrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) between the two groups (Nimenrix+Boostrix Group minus Boostrix Group), in terms of percentage of subjects with anti-T concentrations ≥ 1.0 IU/mL, being greater than or equal to (≥) the pre-defined limit of -10%; Difference in percentage = -0.44, 95% CI 2-sided [-2.48 to 1.26]

3. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: The antibody concentrations were tabulated as adjusted geometric mean concentrations (GMCs) and expressed as international units per millilitre (IU/mL). The primary outcome results only refer to Nimenrix+Boostrix Group and Boostrix Group
Time Frame: One month after Boostrix vaccination (i.e. Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Boostrix Group | Boostrix Group
Number analyzed (Participants) | 225 | 223
IU/mL
  Anti-PT: number analyzed (Participants) | 222 | 223
  Anti-PT | 53.6 [47.2 to 60.8] | 68.0 [59.9 to 77.3]
  Anti-FHA | 316.9 [288.0 to 348.6] | 545.0 [493.2 to 602.4]
  Anti-PRN: number analyzed (Participants) | 224 | 221
  Anti-PRN | 348.3 [293.8 to 412.9] | 499.0 [419.4 to 593.6]
Statistical Analysis 1: Comparison: Nimenrix + Boostrix Group vs Boostrix Group; To demonstrate the non-inferiority of Boostrix co-administered with Nimenrix (Nimenrix+Boostrix Group) compared to Boostrix administered alone (Boostrix Group) with respect to geometric mean concentrations (GMCs) of antibodies against pertussis toxoid (PT), one month after Boostrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) between the two groups (Nimenrix+Boostrix Group minus Boostrix Group) for GMC ratios of antibodies against the pertussis (PT) antigen, being greater than or equal to (≥) the predefined limit of 0.67; ANCOVA; Adjusted GMC ratio = 0.76, 95% CI 2-sided [0.66 to 0.89]
Statistical Analysis 2: Comparison: Nimenrix + Boostrix Group vs Boostrix Group; To demonstrate the non-inferiority of Boostrix co-administered with Nimenrix (Nimenrix+Boostrix Group) compared to Boostrix administered alone (Boostrix Group) with respect to geometric mean concentrations (GMCs) of antibodies against filamentous haemagglutinin (FHA), one month after Boostrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) between the two groups (Nimenrix+Boostrix Group minus Boostrix Group) for GMC ratios of antibodies against the filamentous haemagglutinin (FHA) antigen, being greater than or equal to (≥) the predefined limit of 0.67; ANCOVA; Adjusted GMC ratio = 0.57, 95% CI 2-sided [0.50 to 0.65]
Statistical Analysis 3: Comparison: Nimenrix + Boostrix Group vs Boostrix Group; To demonstrate the non-inferiority of Boostrix co-administered with Nimenrix (Nimenrix+Boostrix Group) compared to Boostrix administered alone (Boostrix Group) with respect to geometric mean concentrations (GMCs) of antibodies against pertactin (PRN), one month after Boostrix vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) between the two groups (Nimenrix+Boostrix Group minus Boostrix Group) for GMC ratios of antibodies against the pertactin (PRN) antigen, being greater than or equal to (≥) the predefined limit of 0.67; ANCOVA; Adjusted GMC ratio = 0.72, 95% CI 2-sided [0.59 to 0.88]

4. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titres Above the Cut-off Values
Description: The reference cut-off values of the assay were rSBA-Men antibody concentrations ≥ 1:128 and ≥ 1:8.
Time Frame: Prior to (i.e. Month 0 for Nimenrix+Boostrix and Nimenrix Groups and Month 1 for Boostrix Group) and one month after Nimenrix vaccination (i.e. Month 1 for Nimenrix+Boostrix and Nimenrix Groups and Month 2 for Boostrix Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 226 | 222 | 223
Participants
  rSBA-MenA ≥ 1:128 | 48 | 46 | 33
  rSBA-MenC ≥ 1:128: number analyzed (Participants) | 225 | 222 | 223
  rSBA-MenC ≥ 1:128 | 224 | 220 | 220
  rSBA-MenW-135 ≥ 1:128 | 13 | 33 | 30
  rSBA-MenY ≥ 1:128 | 225 | 218 | 220
  rSBA-MenA ≥ 1:8 | 31 | 29 | 23
  rSBA-MenC ≥ 1:8 | 226 | 220 | 216
  rSBA-MenW-135 ≥ 1:8 | 80 | 56 | 70
  rSBA-MenY ≥ 1:8 | 226 | 219 | 222

5. Secondary Outcome: Vaccine Response for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibodies
Description: rSBA vaccine response for serogroups A, C, W-135 and Y was defined as:
  * For initially seronegative subjects (pre-vaccination titer below the cut-off of 1:8): number of subjects with rSBA antibody titers ≥ 1:32 one month after vaccination.
  * For initially seropositive subjects (pre-vaccination titer ≥ 1:8): number of subjects with rSBA antibody titers at least four times the pre-vaccination antibody titers, one month after vaccination.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 226 | 222 | 223
Participants
  rSBA-MenA: number analyzed (Participants) | 225 | 222 | 223
  rSBA-MenA | 217 | 207 | 214
  rSBA-MenC | 225 | 210 | 215
  rSBA-MenW-135 | 225 | 216 | 211
  rSBA-MenY | 220 | 214 | 212

6. Secondary Outcome: Anti-D Antibody Concentrations
Description: The antibody concentrations were tabulated as geometric mean concentrations (GMCs) and expressed as international units per milliliter (IU/mL).
Time Frame: Prior to (PRE i.e. Month 0 for Nimenrix + Boostrix Group and Boostrix Group and Month 1 for Nimenrix Group) and one month after Boostrix vaccination (POST i.e. Month 1 for Nimenrix + Boostrix Group and Boostrix Group and Month 2 for Nimenrix Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 225 | 220 | 223
IU/mL
  Anti-D, PRE: number analyzed (Participants) | 217 | 220 | 218
  Anti-D, PRE | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.4]
  Anti-D, POST | 4.0 [3.4 to 4.6] | 4.6 [3.9 to 5.4] | 4.7 [4.0 to 5.4]

7. Secondary Outcome: Anti-T Antibody Concentrations
Description: as for outcome 6
Time Frame: Prior to (i.e. Month 0 for Nimenrix + Boostrix Group and Boostrix Group and Month 1 for Nimenrix Group), one month after Nimenrix vaccination and one month after Boostrix vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 225 | 222 | 223
IU/mL
  Anti-T, pre-vaccination: number analyzed (Participants) | 222 | 222 | 223
  Anti-T, pre-vaccination | 0.6 [0.5 to 0.8] | 0.6 [0.5 to 0.7] | 0.7 [0.5 to 0.8]
  Anti-T, Month 1 | 23.5 [20.8 to 26.5] | 18.5 [16.0 to 21.3] | 13.5 [12.3 to 14.8]
  Anti-T, Month 2: number analyzed (Participants) | 0 | 220 | 223
  Anti-T, Month 2 |  | 13.0 [11.7 to 14.5] | 16.3 [14.6 to 18.2]

8. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations Above the Cut-off Value
Description: The reference cut-off value of the assay was an antibody concentration ≥ 5.0 ELISA units per milliliter (EL.U/mL)
Time Frame: Prior to (i.e. Month 0 for Nimenrix + Boostrix Group and Boostrix Group and Month 1 for Nimenrix Group) and one month after Boostrix vaccination (i.e. Month 1 for Nimenrix + Boostrix Group and Boostrix Group and Month 2 for Nimenrix Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Nimenri+ Boostrix Group: Healthy male or female subjects, between and including 11 and 25 years of age, who received one dose of Nimenrix vaccine co-administered with one dose of Boostrix vaccine, at Month 0, administered by intramuscular injection into the deltoid muscle.
Arm/Group | Nimenri+ Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 225 | 222 | 223
Participants
  Anti-PT, PRE: number analyzed (Participants) | 223 | 222 | 221
  Anti-PT, PRE | 162 | 156 | 153
  Anti-PT, Month 1/Month 2: number analyzed (Participants) | 225 | 220 | 223
  Anti-PT, Month 1/Month 2 | 221 | 220 | 223
  Anti-FHA, PRE: number analyzed (Participants) | 223 | 222 | 223
  Anti-FHA, PRE | 222 | 221 | 220
  Anti-FHA, Month 1/Month 2: number analyzed (Participants) | 225 | 220 | 223
  Anti-FHA, Month 1/Month 2 | 225 | 220 | 223
  Anti-PRN, PRE: number analyzed (Participants) | 223 | 222 | 221
  Anti-PRN, PRE | 200 | 200 | 207
  Anti-PRN, Month 1/Month 2: number analyzed (Participants) | 224 | 218 | 221
  Anti-PRN, Month 1/Month 2 | 223 | 218 | 221

9. Secondary Outcome: Booster Responses for Anti-PT, Anti-FHA and Anti-PRN Concentrations
Description: Booster response to the pertussis components is defined as:
  * For initially seronegative subjects, antibody concentration ≥ 4*cut_off (IU/mL) at one month post-vaccination;
  * For initially seropositive subjects with pre-vaccination antibody concentration < 4*cut_off (IU/mL) : antibody concentration at one month post-vaccination ≥ 4 fold the pre-vaccination antibody concentration;
  * For initially seropositive subjects with pre-vaccination antibody concentration ≥ 4*cut_off (IU/mL) : antibody concentration at one month post-vaccination ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: One month after Boostrix vaccination (i.e. Month 1 for Nimenrix + Boostrix Group and Boostrix Group and Month 2 for Nimenrix Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 222 | 220 | 223
Participants
  Anti-PT antibody (assay cut-off=2.693 IU/mL): number analyzed (Participants) | 222 | 220 | 221
  Anti-PT antibody (assay cut-off=2.693 IU/mL) | 201 | 188 | 201
  Anti-FHA antibody (assay cut-off=2.046 IU/mL) | 208 | 210 | 213
  Anti-PRN antibody (assay cut-off=2.187 IU/mL): number analyzed (Participants) | 221 | 218 | 219
  Anti-PRN antibody (assay cut-off=2.187 IU/mL) | 209 | 198 | 207

10. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Results are presented across doses, after each vaccination (with Nimenrix, Boostrix, total).
Time Frame: During the 4-day (Days 0-3) following each vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 231 | 228 | 232
Participants
  Any Pain, Total | 176 | 148 | 167
  Grade 3 Pain, Total | 15 | 19 | 8
  Any Redness, Total | 81 | 75 | 76
  Grade 3 Redness, Total | 4 | 10 | 6
  Any Swelling, Total | 71 | 71 | 68
  Grade 3 Swelling, Total | 5 | 9 | 7
  Any Pain, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Any Pain, post-Nimenrix | 155 | 121 | 156
  Grade 3 Pain, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Grade 3 Pain, post-Nimenrix | 13 | 12 | 8
  Any Redness, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Any Redness, post-Nimenrix | 64 | 56 | 65
  Grade 3 Redness, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Grade 3 Redness, post-Nimenrix | 3 | 5 | 5
  Any Swelling, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Any Swelling, post-Nimenrix | 57 | 51 | 54
  Grade 3 Swelling, post-Nimenrix: number analyzed (Participants) | 231 | 225 | 232
  Grade 3 Swelling, post-Nimenrix | 3 | 4 | 7
  Any Pain, post-Boostrix | 121 | 101 | 92
  Grade 3 Pain, post-Boostrix | 7 | 8 | 0
  Any Redness, post-Boostrix | 61 | 54 | 39
  Grade 3 Redness, post-Boostrix | 1 | 6 | 4
  Any Swelling, post-Boostrix | 48 | 47 | 33
  Grade 3 Swelling, post-Boostrix | 3 | 5 | 1

11. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination. Results are presented across doses.
Time Frame: During the 4-day (Days 0-3) period following each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 231 | 228 | 232
Participants
  Any Fatigue | 75 | 77 | 81
  Grade 3 Fatigue | 2 | 5 | 4
  Related Fatigue | 70 | 67 | 70
  Any Gastrointestinal symptoms | 23 | 31 | 25
  Grade 3 Gastrointestinal symptoms | 2 | 2 | 1
  Related Gastrointestinal symptoms | 20 | 25 | 18
  Any Headache | 51 | 76 | 65
  Grade 3 Headache | 2 | 5 | 2
  Related Headache | 49 | 67 | 53
  Any Temperature | 14 | 17 | 11
  Grade 3 Temperature | 0 | 0 | 0
  Related Temperature | 10 | 15 | 9

12. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Throughout the study (Month 0 up to Month 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 231 | 228 | 232
Participants | 1 | 5 | 3

13. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events AE(s)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 231 | 228 | 232
Participants | 36 | 44 | 58

14. Secondary Outcome: Number of Subjects With Serious Adverse Events SAE(s)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the study (Month 0 up to Month 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Boostrix Group | Nimenrix Group | Boostrix Group
Number analyzed (Participants) | 231 | 228 | 232
Participants | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) period following each vaccination; Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: throughout the study (Month 0 - Month 2).
Arm/Group | Nimenrix+ Boostrix Group | Nimenrix Group | Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/228 | 0/232
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/228 | 3/232
Other Adverse Events (participants affected / at risk) | 190/231 | 166/228 | 180/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix+ Boostrix Group (N=231) | Nimenrix Group (N=228) | Boostrix Group (N=232)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix+ Boostrix Group (N=231) | Nimenrix Group (N=228) | Boostrix Group (N=232)
Erythema (Skin and subcutaneous tissue disorders) | 81 (81) | 75 (110) | 76 (104)
Fatigue (General disorders) | 75 (75) | 77 (108) | 81 (110)
Gastrointestinal disorder (Gastrointestinal disorders) | 23 (23) | 31 (36) | 25 (28)
Headache (Nervous system disorders) | 54 (54) | 78 (94) | 67 (84)
Nasopharyngitis (Infections and infestations) | 6 (6) | 8 (8) | 15 (16)
Pain (General disorders) | 176 (176) | 148 (222) | 167 (248)
Pyrexia (General disorders) | 15 (15) | 17 (18) | 11 (12)
Swelling (General disorders) | 71 (71) | 71 (98) | 68 (87)

LIMITATIONS AND CAVEATS:
Due to late availability of the serology results, only safety results were posted by the initial due date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.